CLINICAL TRIAL: NCT01041365
Title: Serum 25-hydroxyvitamin D, Vascular Functioning, and Insulin Sensitivity in Adolescent Girls [The DIVA Study (Vitamin D, Insulin, and Vascular Associations)] (Pediatric Physician Training in Translational Research)
Brief Title: Vitamin D, Insulin Sensitivity, and Vascular Associations in Adolescents
Acronym: DIVA
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ambika Ashraf, M.D., Associate Professor, Pediatrics, University of Alabama at Birmingham
Other Study IDs: F090824002
Record Dates: First submitted 2009-12-28; First posted 2009-12-31 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Insulin Sensitivity; Flow-mediated Dilation; Arterial Stiffness
Keywords: insulin sensitivity; vascular function; flow-mediated dilation; arterial stiffness; ethnicity; adolescents; females; glucose tolerance; diabetes; hypertension; cardiovascular
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy adolescents: Healthy adolescent African American and Caucasian females, ages 14-18

SUMMARY:
The overall objectives of this study are to examine the relationships between circulating vitamin D, insulin sensitivity, and multiple indices of vascular function and to examine whether vitamin D deficiency in AA is responsible for ethnic differences in insulin sensitivity and hypertension in AA and EA, as well as mechanisms underlying the association between insulin resistance and blood pressure. We hypothesize that 1) serum 25(OH)D is associated with insulin sensitivity and vascular functioning, independent of adiposity, 2) lower insulin sensitivity and vascular functioning in AA relative to EA is due to lower circulating 25(OH)D in AA, and 3) the relationship between insulin resistance and vascular dysfunction is mediated by 25(OH)D.

Acronyms: African American (AA), European American (EA), Serum 25-hydroxy vitamin D (25()H)D, Body mass index (BMI), Alabama (AL).

ELIGIBILITY:
Inclusion Criteria:

* African American or Caucasian ethnicity
* Ages 14-18 yrs
* Healthy

Exclusion Criteria:

* BMI-for age and -sex higher than 95th centile on the Centers for Disease Control and Prevention Growth Charts
* Use of medication(s) known to influence body composition, vascular function, or glucose metabolism
* Pregnancy
* Diabetes or any chronic diseases

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy adolescent African American and European American teenagers, ages 14-18, will be recruited form the Birmingham, AL community
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | Cross sectional study: at the first study visit

SECONDARY OUTCOMES:
Vascular Function | Cross sectional study: at the second study visit, within 2 weeks of first study visit

CONTACTS AND LOCATIONS:
Overall Officials: Ambika Ashraf, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Ashraf AP, Huisingh C, Alvarez JA, Wang X, Gower BA. Insulin resistance indices are inversely associated with vitamin D binding protein concentrations. J Clin Endocrinol Metab. 2014 Jan;99(1):178-83. doi: 10.1210/jc.2013-2452. Epub 2013 Dec 20. PMID 24170105
- [Derived] Alvarez JA, Gower BA, Calhoun DA, Judd SE, Dong Y, Dudenbostel T, Scholl J, Ashraf AP. Serum 25-hydroxyvitamin D and Ethnic Differences in Arterial Stiffness and Endothelial Function. J Clin Med Res. 2012 Jun;4(3):197-205. doi: 10.4021/jocmr965w. Epub 2012 May 15. PMID 22719806